CLINICAL TRIAL: NCT03094286
Title: A Phase II Exploratory Study of Durvalumab (MEDI4736) in HIV-1 Patients With Advanced Solid Tumors.
Brief Title: Durvalumab in HIV-1 Patients With Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 16/04_DURVAST
Record Dates: First submitted 2017-03-10; First posted 2017-03-29 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: HIV; Cancer
Keywords: HIV; HIV with cancer patient; D006678
MeSH Terms: conditions — Neoplasms | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Durvalumab will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous(IV) administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Durvalumab (MEDI4736) monotherapy at the recommended dose of 1500mg every 4 weeks in solid tumors in HIV-1-infected patients
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab monotherapy of 1500mg every 4 weeks in solid tumors in HIV-1-infected patients until progression significant clinical deterioration, unacceptable toxicity, any criterion for withdrawal from the trial or trial drug is fulfilled
  Other Names: MEDI4736

SUMMARY:
The proposal is a phase II clinical study designed to assess the feasibility of durvalumab (MEDI4736) in HIV-1-infected individuals with solid tumors. Additionally, to obtain data that lets understand the possible benefit of this treatment in cancer patients and HIV infection, exploring if activity of durvalumab (MEDI4736) could be higher in cancer that has been produced at least in part due to the chronic immunosupression. Simultaneously, it will allow us to investigate the effect of disrupting this immunoregulatory pathway might have in reversing cancer pathways and HIV-specific T-cell function during persistent chronic HIV infection in humans.

DETAILED DESCRIPTION:
PD-1/ PD-L1 coinhibitory pathway plays a significant role in the regulation of the immune response in both chronic infectious diseases and cancer.

Preclinical and animal data support the safety and promising activity of anti-PD-1 antibody in HIV-1 infection.

Demonstrated anticancer activity and safety profile of durvalumab (MEDI4736) in cancer clinical trials.

Unlikely drug interactions of durvalumab (MEDI4736) and antiretroviral treatments.

The proposal is a phase II clinical study designed to assess the feasibility of durvalumab (MEDI4736) in HIV-1-infected individuals with solid tumors. Additionally, to obtain data that lets understand the possible benefit of this treatment in cancer patients and HIV infection, exploring if activity of durvalumab (MEDI4736) could be higher in cancer that has been produced at least in part due to the chronic immunosupression. Simultaneously, it will allow us to investigate the effect of disrupting this immunoregulatory pathway might have in reversing cancer pathways and HIV-specific T-cell function during persistent chronic HIV infection in humans.

In this regard, our hypothesis is:

HIV patients with cancer have a similar outcome in terms of tolerability when treated with durvalumab (MEDI4736) monotherapy at the recommended dose than non HIV infected patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age > 18 years at time of study entry.
3. Eastern Cooperative Oncology Group (ECOG) 0-2
4. Life expectancy of > 16 weeks
5. Adequate normal organ and marrow function.
6. Female subjects must either be of non-reproductive potential
7. Subject is willing and able to comply with the protocol
8. Subjects with histologically or cytologically advanced/metatasic-documented lung cancer, head and neck cancer, cervical cancer, melanoma, anal cancer, pancreatic cancer, gastrio-esophageal cancer, triple negative breast cancer, bladder or renal cancer, Cholangiocarcinoma, Kaposi sarcoma, lymphomas, ovarian cancer or Merkel cell carcinoma or any other tumor type in which anti PD-L1 antibodies have desmonstrated antitumoral activity, refractory to standard treatment, intolerant of standard treatment, or for which no standard therapy exists or who refuse the standard treatment.
9. Subjects may be included irrespectively of number of previous lines of treatment for advanced disease.
10. Prior palliative radiotherapy must have been completed at least 2 weeks prior to start the study treatment (subjects may receive localized palliative radiotherapy while receiving study drug).
11. Documented HIV-1 infection.
12. Undetectable viral load in the last analysis.
13. Subjects with brain metastases are eligible if they are asymptomatic, are treated or are neurological stable for at least 2 weeks without the use of steroids or on stable or decreasing dose of<10mb daily prednisone or equivalent.
14. Subjects must be following an antiretroviral therapy at the moment of the inclusion.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study. Previous enrollment in the present study.
2. Participation in another clinical study within last 4 weeks.
3. Other untreated coexisting HIV related malignancies.
4. Any previous treatment with a PD1, PD-L1 or PD-L2 inhibitor, including durvalumab.
5. Receipt of the last dose of anti-cancer therapy within 28 days prior to the first dose of study drug.
6. Mean QT interval corrected for heart rate (QTc) ≥470 ms
7. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab,
8. Any unresolved toxicity (CTCAE grade 2) from previous anti-cancer therapy.
9. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
10. Active or prior documented autoimmune disease within the past 2 years
11. Any syndrome that requires systemic corticosteroid/immunosuppressive medications
12. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
13. History of primary immunodeficiency.
14. History of allogeneic organ transplant.
15. History of hypersensitivity to durvalumab or any excipient.
16. Uncontrolled intercurrent illness
17. Known history of active tuberculosis.
18. Any serious or uncontrolled medical disorder or active infection non HIV, that would impair the ability of the subject to receive the treatment of protocol therapy under treating physician criteria.
19. Subjects with previous malignances, are excluded unless a complete remission was achieved at least 5 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
20. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab.
21. Female subjects who are pregnant, breast-feeding, male, or female patients of reproductive potential who are not employing an effective method of birth control.
22. Symptomatic or uncontrolled brain metastases
23. Subjects with uncontrolled seizures.
24. Patients with tumoral disease in the head and neck region, such as peritracheal or periesophageal lymph node involvement,
25. Patients with neuroendocrine tumors of pulmonary origin or pulmonary metastases with evidence of active bleeding
26. Patients with digestive bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: María González-Cao, MD, Principal Investigator — Instituto Oncológico Dr Rosell
Locations (8):
- Spain (8):
  - ICO-Badalona, Badalona, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - H. Clínic i Provincial de Barcelona, Barcelona
  - H. Universitario Quirón Dexeus, Barcelona
  - Hospital Puerta de Hierro, Madrid
  - H. La Paz, Madrid
  - Hospital Virgen del Rocío, Seville
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Cao M, Moran T, Dalmau J, Garcia-Corbacho J, Bracht JWP, Bernabe R, Juan O, de Castro J, Blanco R, Drozdowskyj A, Argilaguet J, Meyerhans A, Blanco J, Prado JG, Carrillo J, Clotet B, Massuti B, Provencio M, Molina-Vila MA, Mayo de Las Casa C, Garzon M, Cao P, Huang CY, Martinez-Picado J, Rosell R. Assessment of the Feasibility and Safety of Durvalumab for Treatment of Solid Tumors in Patients With HIV-1 Infection: The Phase 2 DURVAST Study. JAMA Oncol. 2020 Jul 1;6(7):1063-1067. doi: 10.1001/jamaoncol.2020.0465. PMID 32271353
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org
- See also: Publication of the results of DURVAST study in this article on JAMA Oncology in 2020 — http://www.ncbi.nlm.nih.gov/pubmed/32271353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2017 and July 2018, a total of 20 patients were enrolled in the study from 7 different sites.
Pre-assignment Details: Screening details:
  Histologically advanced/metatasic lung cancer, head and neck cancer, cervical cancer, melanoma, anal cancer, pancreatic cancer, gastrio-esophageal cancer, triple negative breast cancer, bladder or renal cancer, Cholangiocarcinoma, Kaposi sarcoma, lymphomas, ovarian cancer or Merkel cell carcinoma. HIV infection. Undetectable viral load at last test
Groups:
- Experimental Arm: Durvalumab (MEDI4736) monotherapy at the recommended dose of 1500mg every 4 weeks in solid tumors in HIV-1-infected patients
  Durvalumab: Durvalumab monotherapy of 1500mg every 4 weeks in solid tumors in HIV-1-infected patients until progression significant clinical deterioration, unacceptable toxicity, any criterion for withdrawal from the trial or trial drug is fulfilled.
Period: Overall Study
Arm/Group | Experimental Arm
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.50 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Spain | 20
ECOG [Number; unit: participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  participants
    ECOG 0-1 | 19
    ECOG 2 | 1
Smoking status [Number; unit: participants]
  Former smoker | 9
  Never smoker | 2
  Smoker | 9
Type of Cancer [Number; unit: participants]
  Anal | 2
  Bladder | 1
  Melanoma | 2
  NSCLC | 14
  SCLC | 1
LungCancer(Y/N) [Number; unit: participants]
  Yes | 15
  No | 5
Lung cancer type [Number; unit: participants]
  NSCLC EGFR-, ALK- | 14
  SCLC | 1
  Other | 5
NSCLC histology [Number; unit: participants]
  Adenocarcinoma | 8
  Squamous | 3
  NOS/Undifferenciated | 3
  N/A | 6
Metastasis by cancer type [Number; unit: participants]
  Anal | 2
  Bladder | 1
  Melanoma | 2
  NSCLC | 14
  SCLC | 1
Number of metastatic sites [Number; unit: participants]
  One | 5
  Two | 9
  Three | 4
  Five | 2
Basal CD4-count cells/mm3 [Number; unit: participants]
  <200 | 1
  200-350 | 8
  >350 | 11
HIV-1 group transmission [Number; unit: participants]
  Heterosexual individuals | 6
  MSM | 6
  IDUs | 6
  Unknown | 2
Nº of prior systemic therapies [Number; unit: participants]
  None | 8
  One | 4
  Equal or major of Two | 8
Time since cancer diagnosis [Mean (Standard Deviation); unit: years] | 1.80 (2.80)
Time since HIV diagnosis [Mean (Standard Deviation); unit: years] | 17.68 (10.18)
CD4 at baseline [Mean (Standard Deviation); unit: cells/mm^3] | 416.95 (181.27)
Plasma Viral load at baseline [Mean (Standard Deviation); unit: copies/mL] | 25.39 (15.58)
Treatment duration [Mean (Standard Deviation); unit: Month] | 8.73 (11.57)
Time on treatment and PD-L1 [Mean (Standard Deviation); unit: Month] — Population: Distribution of time on treatment (months) by PD-L1 A total of 15 patients has PD-L1 evaluated
  Month
    PD-1 Negative: number analyzed (Participants) | 11
    PD-1 Negative | 5.97 (8.57)
    PD-1 Positive: number analyzed (Participants) | 4
    PD-1 Positive | 13.18 (6.14)
Distribution of time on treatment for patients with Integrase Inhibitors [Mean (Standard Deviation); unit: Months] — Population: Distribution of time on treatment(months) for patients with/without Integrase Inhibitors in total of all population.
  Months
    With Integrase Inhibitors: number analyzed (Participants) | 14
    With Integrase Inhibitors | 10.90 (13.13)
    Without Integrase Inhibitors: number analyzed (Participants) | 6
    Without Integrase Inhibitors | 3.67 (3.99)

OUTCOME MEASURES:

1. Primary Outcome: Best Response During the Treatment Period
Description: To explore the feasibility of durvalumab (MEDI4736) monotherapy at the recommended dose of 1500mg in solid tumors in HIV-1-infected patients The best overall response is a result of a combination of tumor responses in target and nontarget lesions according to Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: From the first dose until last follow up, assessed up to 24 month
Measure: Number; unit: participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 20
participants
  Complete Response | 1
  Partial Response | 3
  Stable disease | 5
  Progression Disease | 7
  Not Evaluated | 4

2. Secondary Outcome: Duration of Response Global
Description: Only patients with best response Stable disease, Partial Response or Complete response during the treatment period are included in the response analysis.
  Duration of response is the time from response (R) to progression/death (P/D).
Time Frame: From the time from first response evaluation to progression or death, assessed up to 24 months.
Population: Applying a Kaplan -Meyer model the median duration of response is estimated for each type of cancer
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 9
Months
  Anal: number analyzed (Participants) | 1
  Anal | 3.78 (0)
  Melanoma: number analyzed (Participants) | 1
  Melanoma | 7.39 (0)
  NSCLC: number analyzed (Participants) | 7
  NSCLC | 3.7 (1.2)

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the length of time from the date of diagnose to the date of the first documented progression of disease. "Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions".A patient who does not progresses neither dies, is censored at the last tumor evaluation where no progression is detected.
Time Frame: From the date of randomization until end of follow up, assessed up to 24 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 20
Months | 2.5 [1.4 to 5.9]

4. Secondary Outcome: Duration of Response- Dolutegravir/ no Dolutegravir
Description: as for outcome 2
Time Frame: From the date of first response until progression or death, assessed up to 24 months.
Population: Kaplan Meier Estimated median duration of response- Dolutegravir/ no Dolutegravir patients
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Experimental Arm
Number analyzed (Participants) | 9
Month
  Dolutegravir: number analyzed (Participants) | 5
  Dolutegravir | 27.4 [3.7 to 40]
  No Dolutegravir: number analyzed (Participants) | 4
  No Dolutegravir | 2.8 [1.2 to 3.8]

5. Secondary Outcome: Duration of Response by Treatment With INSTIs or no INSTIs
Description: Only patients with best response Stable disease, Partial Response or Complete response during the treatment period are included in the response analysis.
  Duration of response is the time from response to progression/death.
Time Frame: From the date of the first response until progression or death, assessed up to 24 months
Population: Descriptive analysis of response duration - INSTIs (Integrase Inhibitors) or no INSTIs (No Integrase Inhibitors) treated patients
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Experimental Arm
Number analyzed (Participants) | 9
Month
  Integrase Inhibitors: number analyzed (Participants) | 6
  Integrase Inhibitors | 11.32 [3.71 to 27.40]
  No Integrase Inhibitors: number analyzed (Participants) | 3
  No Integrase Inhibitors | 2.10 [1.22 to 3.78]

6. Secondary Outcome: OS Analysis by PD-L1
Description: Kaplan Meier method will be used to estimate the survival function. OS will be mesure at 24 months.
Time Frame: OS is defined as the time from the inclusion date to the death, due to any cause. A patient who does not dies, is censored up to 24 months
Population: Kaplan-Meier model- Summary results of OS - Strata PD-L1 patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 15
Months
  PDL-1 negative: number analyzed (Participants) | 11
  PDL-1 negative | 7.4 [1.2 to 16.3]
  PDL-1 positive: number analyzed (Participants) | 4
  PDL-1 positive | 18.9 [17.0 to 25]

7. Secondary Outcome: OS Analysis by Integrase Inhibitors
Description: OS is defined as the time from the inclusion date to the death, due to any cause. A patient who does not dies, is censored at the last contact date up to 24 months.
Time Frame: From the time from the inclusion date to the death, due to any cause. A patient who does not dies, is censored up to 24 months
Population: Kaplan-Meier model- Summary results of OS- Strata Integrase Inhibitors
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 20
Months
  Integrase Inhibitors: number analyzed (Participants) | 14
  Integrase Inhibitors | 11.5 [4.8 to 18.8]
  No Integrase Inhibitors: number analyzed (Participants) | 6
  No Integrase Inhibitors | 6.0 [0.4 to 33.3]

8. Secondary Outcome: OS Analysis by Dolutegravir
Description: OS is defined as the time from the inclusion date to the death, due to any cause. A patient who does not dies, is censored up to 24 months
Time Frame: as for outcome 7
Population: Kaplan-Meier model- Summary results of OS- Strata patients treated with or without Dolutegravir
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Experimental Arm
Number analyzed (Participants) | 20
Month
  Dolutegravir: number analyzed (Participants) | 10
  Dolutegravir | 12.8 [1.0 to 18.8]
  No Dolutegravir: number analyzed (Participants) | 10
  No Dolutegravir | 8.4 [0.4 to 19.1]

9. Secondary Outcome: PFS Analysis by PD-L1
Description: Progression Free Survival defined as the length of time from the date of diagnosis to the date of the first documented progression of disease
Time Frame: PFS is defined as the time from the inclusion date to the progression or death, due to any cause, up to 24 months patient who does not progresses neither dies, is censored at the last tumor evaluation where no progression is detected.
Population: Summary results Strata by PD-L1 results in cancer patients
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Experimental Arm
Number analyzed (Participants) | 15
Month
  Negative PDL-1: number analyzed (Participants) | 11
  Negative PDL-1 | 2.3 [1.2 to 6.2]
  Positive PDL-1: number analyzed (Participants) | 4
  Positive PDL-1 | 5.7 [4.1 to 17.0]

10. Secondary Outcome: PFS Analysis by Integrase Inhibitors
Description: Defined as the length of time from the date of diagnosis to the date of the first documented progression of disease
Time Frame: From the inclusion date to the progression or death, due to any cause, up to 24 months. patient who does not progresses neither dies, is censored at the last tumor evaluation where no progression is detected.
Population: Kaplan-Meier model- Summary results of PFS by the effect of the presence of Integrase Inhibitors
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 20
Months
  Integrase Inhibitors: number analyzed (Participants) | 14
  Integrase Inhibitors | 2.5 [1.4 to 9.6]
  No Integrase Inhibitors: number analyzed (Participants) | 6
  No Integrase Inhibitors | 2.5 [0.4 to 6.2]

11. Secondary Outcome: PFS Analysis by Dolutegravir
Description: PFS is defined as the time from the inclusion date to the progression or death, due to any cause, date.
Time Frame: From the inclusion date to the progression or death, due to any cause, assessed up to 24 months.
Population: Effect of the presence of Dolutegravir, in the PFS in cancer patients
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Experimental Arm
Number analyzed (Participants) | 20
Month
  Dolutegravir: number analyzed (Participants) | 10
  Dolutegravir | 4.2 [1.0 to 17.0]
  No Dolutegravir: number analyzed (Participants) | 10
  No Dolutegravir | 2.3 [0.4 to 4.1]

ADVERSE EVENTS:
Time Frame: 24 month
Description: The severity of AE will be determined using CTCAE version 4.0.3
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 4/20
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=20)
Vascular arterial ischemia (Vascular disorders) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Blood and lymphatic system disorders) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Death NOS (General disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Confusion (Psychiatric disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatic toxicity (Hepatobiliary disorders) | 1 (1)
Lung infection (Infections and infestations) | 5 (5)
Coronavirus infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=20)
Hypotension (Vascular disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Asthenia (General disorders) | 14 (14)
Pain (General disorders) | 12 (12)
Fever (General disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Prostate syndrom (Reproductive system and breast disorders) | 1 (1)
Serum amylase increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Percardial effusion (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Hepatic toxicity (Hepatobiliary disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Seborreic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Lung infection (Infections and infestations) | 4 (4)
Non respiratory infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03094286/Prot_SAP_000.pdf